CLINICAL TRIAL: NCT07287826
Title: Study for Dexamethasone Mouthwash in Lowering Episodes of Oral Mucositis Among Patients With Cancer: The SMILE Study
Brief Title: Using a Steroid Mouthwash to Prevent Mouth Sores During Chemotherapy
Acronym: SMILE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RP-25-033-WH
Record Dates: First submitted 2025-12-01; First posted 2025-12-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Oral Mucositis Due to Chemotherapy
Keywords: oral mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexamethasone Mouthwash Intervention Group (Experimental): Participants in this arm will receive an alcohol-free dexamethasone mouthwash (0.5 mg per 5 mL solution). They will be instructed to swish and spit 10 mL of the mouthwash for 2 minutes, four times daily, beginning in the first week of chemotherapy. Mouthwash use will continue for at least 8 weeks.
  Interventions: Drug: Dexamethasone Mouthwash

INTERVENTIONS:
Drug: Dexamethasone Mouthwash — Participants will use 10 mL of alcohol-free dexamethasone mouthwash (0.5 mg per 5 mL) as a swish-and-spit rinse for 2 minutes, four times per day. Use will begin during the first week of chemotherapy and continue for at least 8 weeks.

SUMMARY:
The goal of this clinical trial is to learn if a steroid mouthwash (dexamethasone) can prevent mouth sores caused by chemotherapy in adults with cancer. The main questions it aims to answer are:

Does using dexamethasone mouthwash before and during chemotherapy lower the chance of getting moderate to severe mouth sores?

Can this approach reduce pain and improve comfort during chemotherapy?

Researchers will compare patients using the mouthwash to a historical group of patients who received similar chemotherapy but did not use the mouthwash, to see if the mouthwash helps prevent mouth sores.

Participants will:

Use a steroid mouthwash (4 times daily) for up to 8 weeks during chemotherapy

Complete a short weekly survey about mouth discomfort during infusion visits

DETAILED DESCRIPTION:
Oral mucositis is a common and painful side effect of chemotherapy, particularly in patients receiving regimens such as anthracyclines and taxanes. It can lead to difficulty eating, drinking, and speaking, and may result in treatment delays or dose reductions. Recent studies suggest that prophylactic use of dexamethasone mouthwash may reduce the incidence and severity of chemotherapy-induced oral mucositis. However, optimal dosing schedules and broader applicability across cancer types remain unclear.

The SMILE Study is a single-arm, prospective clinical trial designed to evaluate the effectiveness of dexamethasone mouthwash in preventing oral mucositis in adults receiving specific types of chemotherapy for cancer. Participants will be enrolled before beginning chemotherapy regimens known to be associated with a high risk of mucositis. All participants will receive dexamethasone mouthwash to use as a swish-and-spit rinse for 8 weeks.

The study will enroll at least 45 participants. Participants will be monitored throughout their chemotherapy treatment for signs and symptoms of oral mucositis, treatment adherence, and potential adverse events related to the mouthwash. Patient-reported outcomes will be collected using the Oral Mucositis Weekly Questionnaire (OMWQ), administered at routine infusion visits. Data on chemotherapy dose modifications or delays will also be recorded.

To assess effectiveness, the outcomes from the prospective cohort will be compared to a retrospective historical control group composed of patients previously treated at the same facility with similar chemotherapy regimens but who did not receive dexamethasone mouthwash. Data from the control group will be collected from the electronic medical record (EMR) and will include oral mucositis incidence and severity, chemotherapy regimens, and any treatment delays due to mucositis. Matching or statistical adjustment methods (e.g., multivariable regression) may be used to account for confounding variables.

The primary endpoint is the incidence of grade ≥2 oral mucositis during chemotherapy, graded per CTCAE v5.0. Secondary endpoints include overall mucositis severity, chemotherapy delays or reductions, patient-reported symptoms (pain, discomfort, interference with eating or speaking), and adherence to mouthwash use.

Risks related to the intervention are expected to be minimal and may include oral thrush, burning sensation, or changes in taste. Dexamethasone is generally well tolerated in topical formulations, and safety monitoring will focus on local and systemic reactions potentially linked to steroid use.

There is no cost to participate in the study. All study activities are conducted as part of routine care at Woman's Cancer Pavilion. The study is funded by a grant from the Foundation for Woman's.

This study will not collect biospecimens. No genetic testing will be performed. Only de-identified data will be used in any publication or external reporting. Identifiable information from the prospective and historical cohorts will be stored securely in compliance with institutional and federal regulations.

This research aims to generate evidence to support proactive, standardized interventions to prevent chemotherapy-induced oral mucositis and improve supportive care for patients undergoing cancer treatment.

ELIGIBILITY:
Inclusion criteria:

* ≥18 years old
* Confirmed cancer diagnosis
* Scheduled to receive or receiving chemotherapy known to be associated with oral mucositis (e.g., anthracyclines and taxanes)
* Ability to provide informed consent
* Ability to comply with study procedures

Exclusion criteria:

* Current tobacco usage or usage within the past 6 weeks.
* HIV/AIDS
* Gastrointestinal disorder (such as Crohn's disease, ulcerative colitis, or celiac disease)
* History of cold sores (herpes simplex virus)
* Herpes zoster (oral shingles) within the past 6 weeks
* Active oral infections at the time of enrollment (e.g., candidiasis)
* Known sensitivity or allergy to dexamethasone
* Inability to self-administer or tolerate mouthwash protocol
* Concurrent enrollment in conflicting clinical trials
* Existing oral ulcers or oral mucositis at enrollment
* Pregnant
* Uncontrolled diabetes mellitus as defined by HbA1c unknown or >8% in the past 3 months despite adequate therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade ≥2 Oral Mucositis | From start of chemotherapy through completion of first chemotherapy cycle (up to 8 weeks)
  Proportion of participants who develop grade 2 or higher oral mucositis, as assessed by Common Terminology Criteria for Adverse Events (CTCAE v5.0), during chemotherapy treatment while using dexamethasone mouthwash.

SECONDARY OUTCOMES:
Severity of Oral Mucositis Symptoms (Clinician Assessed) | From start of chemotherapy through completion of first chemotherapy cycle (up to 8 weeks)
  Severity of oral mucositis will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE v5.0) grading scale.
Severity of Oral Mucositis Symptoms (Patient-Reported) | From start of chemotherapy through completion of chemotherapy cycle 1 (up to 8 weeks)
  Participants will report symptoms using the Oral Mucositis Weekly Questionnaire (OMWQ), which includes ratings for mouth and throat soreness, pain, and interference with eating, drinking, and speaking.
Chemotherapy Treatment Modifications Due to Oral Mucositis | Up to 16 weeks
  Number of chemotherapy dose delays, reductions, or discontinuations that are documented as being caused by oral mucositis symptoms.
Number of Participants With Adverse Events Related to Dexamethasone Mouthwash | Up to 16 weeks
  Number of participants who experience at least one adverse event (AE) deemed related to mouthwash use, including but not limited to oral candidiasis or allergic response.
Mouthwash Adherence | Daily for the first 8 weeks of chemotherapy
  Self-reported and staff-monitored adherence to the prescribed mouthwash use protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jaymes H Collins, PhD, Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time, it is not yet known whether individual participant data (IPD) from this study will be shared. If shared, the IPD may include de-identified data sets containing clinical outcomes such as oral mucositis severity, adverse events, and participant-reported symptom scores. A final decision will be based on privacy protections, data use agreements, and institutional policies related to secondary data sharing.

REFERENCES:
- [Background] Saigal B, Guerra L. Prevention of Stomatitis: Using Dexamethasone-Based Mouthwash to Inhibit Everolimus-Related Stomatitis. Clin J Oncol Nurs. 2018 Apr 1;22(2):211-217. doi: 10.1188/18.CJON.211-217. PMID 29547614
- [Background] Krishnaswamy V. A thin, flat, parallel plate ionization chamber for electron beam depth-dose measurements. Radiology. 1973 Oct;109(1):223-4. doi: 10.1148/109.1.223. No abstract available. PMID 4209263
- [Background] Kuderer NM, Desai A, Lustberg MB, Lyman GH. Mitigating acute chemotherapy-associated adverse events in patients with cancer. Nat Rev Clin Oncol. 2022 Nov;19(11):681-697. doi: 10.1038/s41571-022-00685-3. Epub 2022 Oct 11. PMID 36221000
- [Background] Ruddy KJ, Zahrieh D, He J, Waechter B, Holleran JL, Lewis LD, Chow S, Beumer J, Weiss M, Trikalinos N, Faller B, Lustberg M, Rugo HS, Loprinzi C. Dexamethasone to prevent everolimus-induced stomatitis (Alliance MIST Trial: A221701). Semin Oncol. 2023 Feb-Apr;50(1-2):7-10. doi: 10.1053/j.seminoncol.2023.01.001. Epub 2023 Jan 17. PMID 36693773
- [Background] Kuba S, Maeda S, Shibata K, Soutome S, Yamanouchi K, Matsumoto M, Tanaka A, Morita M, Hatachi T, Otsubo R, Yano H, Kawashita Y, Sato S, Taniguchi H, Kanetaka K, Umeda M, Nagayasu T, Eguchi S. EFFICACY AND SAFETY OF A DEXAMETHASONE-BASED MOUTHWASH TO PREVENT CHEMOTHERAPY-INDUCED STOMATITIS IN WOMEN WITH BREAST CANCER: A MULTICENTRE, OPEN-LABEL, RANDOMISED PHASE 2 STUDY. J Evid Based Dent Pract. 2023 Sep;23(3):101896. doi: 10.1016/j.jebdp.2023.101896. Epub 2023 Jun 11. PMID 37689451
- [Background] Rugo HS, Seneviratne L, Beck JT, Glaspy JA, Peguero JA, Pluard TJ, Dhillon N, Hwang LC, Nangia C, Mayer IA, Meiller TF, Chambers MS, Sweetman RW, Sabo JR, Litton JK. Prevention of everolimus-related stomatitis in women with hormone receptor-positive, HER2-negative metastatic breast cancer using dexamethasone mouthwash (SWISH): a single-arm, phase 2 trial. Lancet Oncol. 2017 May;18(5):654-662. doi: 10.1016/S1470-2045(17)30109-2. Epub 2017 Mar 15. PMID 28314691

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT07287826/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT07287826/ICF_001.pdf